CLINICAL TRIAL: NCT05619575
Title: A Pre-market, Open-label, Within Subject Study, of Acceptance and Performance of the CP1170 Sound Processor in Experienced Adult Cochlear Implant Recipients Compared With the CP1150 Sound Processor and Their Current Sound Processor.
Brief Title: Acceptance and Performance of the CP1170 Sound Processor in Experienced Adult Cochlear Implant Recipients
Acronym: POLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLTD5836
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CP1170 Sound Processor (Experimental): Take home use of CP1170 Sound Processor for 2 weeks followed by in-booth testing of this investigational device. The SCAN 2 FF (automated ForwardFocus On) program will be compared to the SCAN 2 (ForwardFocus Off) program in the CP1170 Sound Processor. This investigational device will also be compared to the CP1150 Sound Processor and participants' own sound processor.
  Interventions: Device: CP1170 Sound Processor; Device: CP1150 Sound Processor

INTERVENTIONS:
Device: CP1170 Sound Processor — The CP1170 Sound Processor will be used to determine the hearing performance with the new implementation of ForwardFocus in SCAN 2 (SCAN 2 FF), as assessed by speech perception in noise.
Device: CP1150 Sound Processor — Active comparator off-the-ear sound processor.

SUMMARY:
Acceptance and performance of the CP1170 sound processor in experienced adult cochlear implant recipients compared with the CP1150 sound processor and their current sound processor.

DETAILED DESCRIPTION:
This investigation is planned to investigate the performance and clinical benefits of features that are new to the CP1170 Sound Processor. This study will build on the evidence previously collected on off-the-ear (OTE) sound processors and ForwardFocus, with particular focus on the acceptance and satisfaction of the automation of ForwardFocus in the CP1170 Sound Processor and associated components in general.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Post lingually deafened
3. Implanted with the CI600 Series (CI612, CI632, CI622, CI624), CI500 Series (CI512, CI532, CI522); Freedom Series (CI24RE(CA), CI24RE(ST), CI422) or N24 Series (CIC3).
4. At least 6 months experience with a cochlear hearing implant
5. At least 3 months experience with any Nucleus sound processor and SCAN program
6. Able to score 30% or more at +15 SNR with CI alone on a sentence in babble test
7. Willingness to participate in and to comply with all requirements of the protocol
8. Fluent speaker in English as determined by the investigator
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Additional disabilities that would prevent participation in evaluations
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedures
3. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling
5. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation, as determined by the Investigator.
6. Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Macquarie, Macquarie, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults With a Cochlear Implant: All study participants (post-lingually deafened adults with at least 6 months experience with a cochlear implant and 3 months experience with SCAN program).
Period: Overall Study
Arm/Group | Adults With a Cochlear Implant
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adults With a Cochlear Implant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 63.4 [35 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Primary Outcome: Paired Difference in dB SRT Between the CP1170 SCAN 2 FF (Automated ForwardFocus ON) and CP1170 SCAN 2 (ForwardFocus OFF) in 65 dB SPL (Sound Pressure Level) S0Nrearhalf 4Talker Babble (Speech Perception in Noise)
Description: Speech perception in noise was measured using the Australian Speech Test In Noise (AUSTIN), which is a test that uses Bamford-Kowal-Bench (BKB)-like target sentences presented in adaptive noise. The goal of the speech perception test in noise was to provide the speech-to-noise ratio for 50% speech intelligibility.
Time Frame: During a Single Ad-Hoc Visit (between Day 141 - Day 218)
Measure: Mean (95% Confidence Interval); unit: dB SRT
Groups:
- All Participants: Participants completed a hearing test using CP1170 with automated ForwardFocus switched on (SCAN 2 FF) or ForwardFocus switched off (SCAN 2).
Arm/Group | All Participants
Number analyzed (Participants) | 17
dB SRT
  CP1170 SCAN 2 FF | -6.58 [-8.38 to -4.77]
  CP1170 SCAN 2 | -4.58 [-6.30 to -2.86]
  Difference between CP1170 SCAN 2 FF and SCAN 2 | -2.00 [-2.82 to -1.18]

2. Secondary Outcome: Paired Difference in dB SRT Between the CP1170 SCAN 2 FF (Automated ForwardFocus ON) and CP1170 SCAN 2 (ForwardFocus OFF) in 65 dB SPL S0N3 Babble (Speech Perception in Noise)
Description: as for outcome 1
Time Frame: During a single Ad-Hoc Visit (anytime between Day 141 - Day 218)
Measure: Mean (95% Confidence Interval); unit: dB SRT
Groups:
- All Participants: Participants completed a hearing test using CP1170 with automated ForwardFocus switched on (SCAN 2 FF) and ForwardFocus switched off (SCAN 2).
Arm/Group | All Participants
Number analyzed (Participants) | 17
dB SRT
  CP1170 SCAN 2 FF | -4.66 [-6.65 to -2.67]
  CP1170 SCAN 2 | -3.24 [-5.29 to -1.18]
  Difference between SCAN 2 FF and SCAN 2 | -1.43 [-2.20 to -0.65]

3. Secondary Outcome: Paired Difference in Percentage CNC (Consonant-nucleus-consonant) Words Correct in Quiet (50 dB) Between the CP1170 Sound Processor and CP1150 Sound Processor (Commercial Version)
Description: Speech perception in quiet was measured using the CNC monosyllabic words at 50 dB SPL from S0 position. The goal of speech perception assessment in quiet was to compare % words correct for each of the conditions.
Time Frame: During Ad-Hoc Visit (anytime between Day 127 - Day 190)
Measure: Mean (95% Confidence Interval); unit: Percentage of correct words
Groups:
- CP1170 Sound Processor: Take home use of CP1170 Sound processor for 2 weeks followed by in booth testing of the investigational device. This was compared to the in booth testing of CP1150 sound processor.
Arm/Group | CP1170 Sound Processor
Number analyzed (Participants) | 17
Percentage of correct words
  CP1170 SCAN 2 | 59.06 [51.91 to 66.21]
  CP1150 SCAN | 56.53 [49.09 to 63.97]
  Difference between CP1170 and CP1150 | 2.53 [-0.41 to 5.47]

4. Secondary Outcome: Subjective Acceptance and Satisfaction Between the CP1170 Sound Processor and the Subject's Own Processor
Description: Number of participants who were somewhat or very satisfied with the overall sound quality of their SCAN program (SCAN in own sound processor, SCAN 2 FF in CP1170) as indicated through two questionnaires. The CP1170 Questionnaire and Baseline Questionnaire have a 5-point Likert scale for each rating (with the values ranging from: 1 = least favourable option to 3 = Neutral to 5 = most favourable option).
Time Frame: 2 weeks
Population: At baseline, 20 participants completed the Baseline Questionnaire. As three participants did not complete the study, the CP1170 Questionnaire was completed by 17 participants rather than 20.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants completed a questionnaire at baseline to provide their subjective ratings on their own sound processor device. Participants then completed a questionnaire after a minimum of two weeks actual use of the CP1170 Sound Processor.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Participants
  CP1170 Sound Processor: number analyzed (Participants) | 17
  CP1170 Sound Processor | 16
  Own Sound Processor | 18

5. Secondary Outcome: Paired Difference in Global SSQ12 Scores After Experience With the CP1170 Sound Processor and Own Processor
Description: The SSQ12, which measures subjective hearing performance, is comprised of 12 items using the response format on a scale from 0 to 10, where 0 equals no ability and 10 equals perfect ability. These are divided into three sub-scales and the questions 1-5 are from the speech sub-scale, 6-8 from the spatial, and 9-12 from the qualities sub-scale. The three sub-scales are the average of the questions within. A 'not applicable' option is given for each item. The change from baseline is then calculated and the theoretical score could vary between -10 to +10. The higher the score, the higher the benefit. A positive score indicates improved hearing, and a negative value indicates impaired hearing.
Time Frame: During a Single Ad-Hoc Visit (anytime between Day 23 - Day 70)
Population: Twenty participants completed the SSQ12 at Baseline for their own sound processor, however, due to subject attrition, only 18 participants completed the questionnaire on the CP1170 Sound Processor.
Measure: Mean (95% Confidence Interval); unit: SSQ12 Global score
Groups:
- All Participants: Participants completed the Speech, Spatial and Qualities of Hearing (SSQ12) scale at baseline to provide their subjective ratings on their own device, and then again after experience with the CP1170 Sound Processor.
Arm/Group | All Participants
Number analyzed (Participants) | 20
SSQ12 Global score
  CP1170 Sound Processor: number analyzed (Participants) | 18
  CP1170 Sound Processor | 6.07 [5.31 to 6.83]
  Own Sound Processor | 6.06 [5.29 to 6.83]
  Difference between CP1170 and own sound processor: number analyzed (Participants) | 18
  Difference between CP1170 and own sound processor | 0.10 [-0.52 to 0.72]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Adults With a Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With a Cochlear Implant (N=20)
Ear-related adverse event (Ear and labyrinth disorders) | 6 (6)
Non ear-related (Gastrointestinal disorders) | 1 (1) — Gastrointestinal problem

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT05619575/Prot_SAP_000.pdf